CLINICAL TRIAL: NCT04581993
Title: Effectiveness of Specialized Nutritious Foods, Social and Behavior Change Communication Interventions to Prevent Stunting Among Children in Badakhshan Province, Afghanistan: a Quasi-experimental Study
Brief Title: Effectiveness of SNF and SBCC to Prevent Stunting Among Children in Afghanistan: a Quasi-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Ministry of public Health Afghanistan (Unknown); United Nations World Food Programme (WFP) (Other); The Aga Khan Foundation (Other); Aga Khan Health Services (Other)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Professor, Aga Khan University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Stunting Study Afghanistan
Record Dates: First submitted 2020-10-08; First posted 2020-10-09 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Stunting; Malnutrition, Child
Keywords: Stunting; Children; Specialized Nutritious Foods; Social and Behavior Change Communication; Afghanistan
MeSH Terms: conditions — Growth Disorders; Child Nutrition Disorders | interventions — Sugars

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Pregnant and lactating women (PLW) will receive Super Cereal - wheat soya blend with sugar and children aged 6-23 months will receive lipid-based nutrient supplement-medium quantity (LNS-MQ). Social and behavior change communication (SBCC), community mobilization, referrals, identification of model families, food demonstrations, local recipe) ration/beneficiary entitlement cards will be provided for easy verification and tracking during delivery of intervention.
  Interventions: Dietary Supplement: Super Cereal - wheat soya blend with sugar; Dietary Supplement: Lipid-based nutrient supplement-medium quantity (LNS-MQ); Behavioral: Social and behavior change communication (SBCC)
- Control (No Intervention): Control districts will receive routine health care services available in the study area.

INTERVENTIONS:
Dietary Supplement: Super Cereal - wheat soya blend with sugar — Pregnant and lactating women will received Super Cereal during pregnancy and first six months of lactation.
  Arms: Intervention
Dietary Supplement: Lipid-based nutrient supplement-medium quantity (LNS-MQ) — Children will receive LNS during 6-23 months of age.
  Arms: Intervention
Behavioral: Social and behavior change communication (SBCC) — SBCC will be provided to improve care-givers knowledge, attitudes and practices related to infant and young child feeding.
  Arms: Intervention

SUMMARY:
Over the years, there has been some progress made in reducing stunting in Afghanistan, the prevalence remains high with half of the provinces experiencing rates above the WHO alert threshold. As part of the Country Strategic Plan (CSP), the World Food Programme (WFP) plans to implement a stunting prevention programme in collaboration with Ministry of Public Health (MoPH) through its Public Nutrition Department (PND) in selected locations with stunting rates above 45%. The programme will emphasis on appropriate nutrition support in the '1000 days' window of opportunity with special focus on proven effective nutrition interventions such appropriate breast feeding, complementary feeding, micronutrient supplementation, malnutrition treatment and prevention, WASH.

DETAILED DESCRIPTION:
Over the years, there has been some progress made in reducing stunting in Afghanistan, the prevalence remains high with half of the provinces experiencing rates above the WHO alert threshold. As part of the Country Strategic Plan (CSP), the World Food Programme (WFP) plans to implement a stunting prevention programme in collaboration with Ministry of Public Health (MoPH) through its Public Nutrition Department (PND) in selected locations with stunting rates above 45%. The programme will emphasis on appropriate nutrition support in the '1000 days' window of opportunity with special focus on proven effective nutrition interventions such appropriate breast feeding, complementary feeding, micronutrient supplementation, malnutrition treatment and prevention, WASH. This will therefore take the form of an integrated approach ensuring the targeted beneficiaries are supported to access nutrition assistance as well as other complimentary interventions provided in-kind by study partners or promoted through social and behaviour change communication (SBCC). WFP will target pregnant and lactating women (PLW) and children aged 6-23 months but will also engage men and players that influence maternal infant and young child nutrition practices. Through this programme, children aged 6-23 months will receive lipid-based nutrient supplement - medium quantity (LNS-MQ) to complement their diets while PLW will receive Super Cereal - wheat soya blend with sugar.

An operational research study was embedded in the stunting prevention programme by credible third-party to determine the extent to which the new actions will influence nutrition outcomes and practices. Introducing the provision of SNF, SBCC as well as formulation and adoption of local culturally acceptable recipes for complementary feeding from locally available nutritious food would be new additions to the current Community Based Nutrition Program (CBNP) package in the implementation phase. During the project implementation, emphasis will be placed will be placed on the adoption of the locally formulated complementary foods as well as application of knowledge and practices promoted through the SBCC activities as part of the exit strategy and ensuring a lasting impact of the project.

Therefore, the Centre of Excellence in Women and Child Health, Aga Khan University, Pakistan proposes an operational research study with mix-methods including formative research, quasi-experimental design to evaluate the stunting prevention programme and process evaluations for stronger evidence base on the effectiveness of proposed interventions on prevention of stunting and developing viable programmes on nutrition under "real" operational conditions.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and lactating women
* Children 6-23 months
* Willing to participate

Exclusion Criteria:

* Non pregnant and lactating women
* Children >24 months
* Refuse to participate

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction in stunting | 18 months
  10% reduction in stunting among children 6-23 months in the intervention compare to control

CONTACTS AND LOCATIONS:
Overall Officials: Sajid B Soofi, MBBS, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan Health Services, Fayzabad, Badakhshān, Afghanistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soofi SB, Khan GN, Sajid M, Hussainyar MA, Shams S, Shaikh M, Ouma C, Azami S, Naeemi M, Hussain A, Umer M, Hussain I, Ahmed I, Ariff S. Specialized nutritious foods and behavior change communication interventions during the first 1000 d of life to prevent stunting: a quasi-experimental study in Afghanistan. Am J Clin Nutr. 2024 Sep;120(3):560-569. doi: 10.1016/j.ajcnut.2024.07.007. Epub 2024 Jul 14. PMID 39004283